CLINICAL TRIAL: NCT02195557
Title: Synvisc® in Knee Osteoarthritis: Retrospective Follow-up in Treated Patients Since at Least Three Years
Brief Title: Retrospective Follow-up Study of Synvisc® in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1139.6
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — hylan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Synvisc®
  Interventions: Drug: Synvisc®

INTERVENTIONS:
Drug: Synvisc®

SUMMARY:
Retrospective collection of data, aimed at a better knowledge of the use of Synvisc® among the patients with knee osteoarthritis (OA) since at least three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee osteoarthritis using Synvisc® since at least three years

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: rheumatological practice
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2002-04; Primary Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Reason for prescription | at least 3 years before start of observation period
Number of other treatments per patient | at least 3 years of observation
  antalgics, non-steroid anti-inflammatory drugs (NSAIDs), steroid anti-inflammatory drugs (SAIDs), specific symptomatic treatments and surgery
Time between two treatments | at least 3 years of observation